CLINICAL TRIAL: NCT06453564
Title: Cross Validation of Body Composition Measurement
Status: Enrolling by invitation | Type: Observational
Sponsor: John R. Speakman (Other)
Responsible Party: Sponsor-Investigator, John R. Speakman, Principal Investigator, Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Organization: Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences (Other)
Other Study IDs: SIAT-IRB-221115-H0630
Record Dates: First submitted 2024-04-17; First posted 2024-06-11 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Body Composition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 18.5≤ BMI <23.9: The investigators planned to recruit 10 volunteers with a BMI between 18 and 23. Half male, half female. There are no age restrictions. Because there are large differences in body composition among people with different BMI, there are also differences between men and women. The investigators will look at the differences in body composition measured by different methods for each individual in this group.
- 24≤BMI<27.9: The investigators planned to recruit 10 volunteers with a BMI between 23 and 30. Half male, half female. There are no age restrictions. The volunteers in this group were relatively underweight. The investigators will look at the differences in body composition measured by different methods for each individual in this group.
- 28≤BMI<35: The investigators planned to recruit 10 volunteers with a BMI between 30 and 35. Half male, half female. There are no age restrictions. The volunteers in this group were obese patients. The investigators will look at the differences in body composition measured by different methods for each individual in this group.

SUMMARY:
Obesity, as a chronic disease, has emerged as one of the most pressing health concerns in the 21st century. According to statistics, over 2.1 billion individuals worldwide are affected by overweight or obesity. It is worth noting that obesity ranks fifth among the leading causes of mortality globally. Body fat percentage (fat%) serves as an accurate measure for evaluating body fat content, which can be further categorized into subcutaneous fat, intra-abdominal fat, and intra-organ fat. Subcutaneous fat primarily functions in heat preservation and energy storage while intra-abdominal fat plays a crucial role in safeguarding internal organs from harm. Visceral fat deposition mainly occurs due to intracellular lipid degeneration within organ cells. Extensive research has demonstrated significant variations in metabolic indications and risks associated with different types of fats across various body regions. Therefore, precise segmentation and quantification of overall body fat composition and its distribution hold immense significance for studying individual obesity characteristics, predicting health outcomes, facilitating clinical diagnosis, and devising effective treatment strategies. However, it should be noted that current instruments used for measuring body composition exhibit varying levels of accuracy. Henceforth, this study aims to cross-validate several commonly employed body composition analyzers including DXA (Dual-energy X-ray Absorptiometry), BIA (Bioelectrical Impedance Analysis), BODPOD (Air Displacement Plethysmography), MRI (Magnetic Resonance Imaging), deuterium dilution technique, and 3D laser scanning techniques to assess their agreement and discrepancies when measuring different aspects of body composition.

DETAILED DESCRIPTION:
Cross validation of body composition measurement

Body composition will be measured by the following methods:

The fasting body weight and height were measured using the Seca medical metric system (Seca 311231, Germany). Volunteers were instructed to wear a standardized disposable lab coat and stand barefoot on an electronic scale for accurate measurements. Barefoot height was measured to the nearest millimeter using a commercially available Leicester stadiometer (Seca 217, Germany). Volunteers were positioned in the center of the 3D scanning room (Scanatic™ 360) and instructed to maintain proper posture while our scanning staff operated the scanner, sensor, and camera in order to obtain precise human dimensional data including waist circumference and hip circumference.

BIA (Bioelectrical Impedance Analysis):

The TANITA device (TANITA- mc980) provides individual weight measurements for the right arm, left arm, trunk, right leg, and left leg. Additionally, it generates a comprehensive body composition report that includes body weight (BW), percentage of body fat (fat%), body fat mass (FM), BMI, and fat-free mass (FFM).

DXA (Dual-energy X-ray Absorptiometry):

During DXA measurements (Horizon, Hologic), all volunteers will be required to wear uniform disposable lab coats and remove any metal accessories. Dual-energy X-ray absorptiometry (DXA) utilizes a low dose X-ray beam with two energy peaks, one predominantly absorbed by soft tissues and the other mainly absorbed by bone, to assess the whole body at the workbench. This enables quick differentiation of bone fraction from total body composition and provides penetration analysis of soft tissue through software algorithms for accurate determination of fat mass and fat-free mass.

BODPOD (Air Displacement Plethysmography):

Prior to the test, the volunteers underwent a fasting period and refrained from engaging in exercise, intense physical activity, or smoking within two hours. To minimize any potential impact on measurement results, it was required for them to wear a well-fitting swimsuit (boxers for men; one-piece bathing suit for women), a swimming cap, and remove all accessories (such as watches, necklaces, earrings, rings, and socks) from their bodies. BODPOD (GS-X, Cosmed) operates on the principle of air displacement similar to the classical underwater weighing method. Utilizing a 2-component model approach based on body composition analysis divides it into two components: body fat and free fat mass. By measuring gas volume displaced and considering differences in density between fat and non-fat tissues along with volunteer's body weight data upon entering the test chamber allows calculation of both percentage of body fat and percentage of lost body fat.

MRI (Magnetic Resonance Imaging):

This experiment used cutting-edge magnetic resonance imaging (MRI, United-Imaging Healthcare, uMR790) instrument measurement, no injection of contrast medium, volunteers lie flat on the MRI bed body, using a newly developed rapid magnetic resonance dynamic imaging sequence to scan the whole body covering the neck to the knee, MRI scanning by trained professionals. All subjects will undergo the test, and the data collected will be used to assist in the development of computer language programming for whole-body fat quantification and segmentation.

Deuterium dilution technology:

Over the past 50 years, stable isotope technology has been extensively utilized in the field of human nutrition. Deuterium, a stable and nonradioactive isotope of hydrogen, is employed in the form of deuterium oxide which is orally administered to volunteers and thoroughly mixed with their body water. Subsequently, it is excreted through urine, saliva, sweat, and milk. The recycling process of deuterium oxide within the body mirrors that of regular water as it becomes dispersed throughout the body and eventually expelled. This technique can be applied to both adults and children; moreover, by providing lactating mothers with deuterium oxide water intake data can be obtained regarding breast milk consumption by breastfed infants. Prior to administering water, baseline urine samples were collected from adult participants who then received 30g of precisely measured deuterated oxide water (with an accuracy up to 0.001g). Three hours later, additional urine samples were collected for analysis purposes. By examining changes in deuterium abundance within these samples, calculations can be made regarding total body water content while fat weight can be determined using the formula FFM(kg) = TBW (kg)/0.732.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* BMI ranges between 18-35 kg/m2

Exclusion Criteria:

* current pregnancy or pregnancy within the last 12 months, and/or currently breast feeding or lactating
* Individuals with known non-communicable disease notably diabetes, cardiovascular disease or cancer
* any diseases or chronic use of medications that would influence ability to comply with the study requirements

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population was healthy. The women were not pregnant or planning to become pregnant and were lactating. None of the volunteers had metal implants in their bodies. All volunteers had no serious metabolic diseases that would affect the trial.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2026-07-19 (Estimated); Study Completion 2026-07-19 (Estimated)

PRIMARY OUTCOMES:
Weight | About 10 minutes.
  Weight in kilograms will be measured by scale (Seca 311231, Germany), DXA (Dual-energy X-ray Absorptiometry), TANITA, BODPOD (Air Displacement Plethysmography).
Height | About 5 minutes.
  Height in centimetres will be measured by Leicester stadiometer(Seca 217, Germany).
BMI | About 10 minutes (calculated).
  BMI values in kg/m2 were calculated from weight measured by TANITA and height measured by Leicester stadiometer (Seca 217, Germany).
Fat mass | About two weeks (including the time to calculate the MIR results).
  Fat mass in kilograms will be measured by DXA (Dual-energy X-ray Absorptiometry), TANITA, MRI (United imaging uMR790 and BODPOD (Air Displacement Plethysmography). Total body fat in cubic centimeters will be converted to fat mass in kilograms using body density.
Fat free mass | About three weeks (including the sample analysis time taken by the deuterium dilution technique).
  Fat mass in kilograms will be measured by DXA (Dual-energy X-ray Absorptiometry), TANITA, BODPOD (Air Displacement Plethysmography) and deuterium dilution method.
Fat% | About two weeks (including the time to calculate the MIR results).
  Fat% will be measured by DXA (Dual-energy X-ray Absorptiometry), TANITA, BODPOD (Air Displacement Plethysmography) and MRI (United imaging uMR790).
Total body water | About three weeks (including the sample analysis time taken by the deuterium dilution technique).
  Total body water in kilograms will be measured by TANITA and deuterium dilution method.
Total body volume | About a week.
  Total body volume in liters will be measured by BODPOD (Air Displacement Plethysmography) and MRI (United imaging uMR790).

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Institutes of advanced technology, Shenzhen, Guangdong, China

REFERENCES:
- [Background] Speakman JR, Yamada Y, Sagayama H, Berman ESF, Ainslie PN, Andersen LF, Anderson LJ, Arab L, Baddou I, Bedu-Addo K, Blaak EE, Blanc S, Bonomi AG, Bouten CVC, Bovet P, Buchowski MS, Butte NF, Camps SGJA, Close GL, Cooper JA, Creasy SA, Das SK, Cooper R, Dugas LR, Ebbeling CB, Ekelund U, Entringer S, Forrester T, Fudge BW, Goris AH, Gurven M, Hambly C, El Hamdouchi A, Hoos MB, Hu S, Joonas N, Joosen AM, Katzmarzyk P, Kempen KP, Kimura M, Kraus WE, Kushner RF, Lambert EV, Leonard WR, Lessan N, Ludwig DS, Martin CK, Medin AC, Meijer EP, Morehen JC, Morton JP, Neuhouser ML, Nicklas TA, Ojiambo RM, Pietilainen KH, Pitsiladis YP, Plange-Rhule J, Plasqui G, Prentice RL, Rabinovich RA, Racette SB, Raichlen DA, Ravussin E, Reynolds RM, Roberts SB, Schuit AJ, Sjodin AM, Stice E, Urlacher SS, Valenti G, Van Etten LM, Van Mil EA, Wells JCK, Wilson G, Wood BM, Yanovski J, Yoshida T, Zhang X, Murphy-Alford AJ, Loechl CU, Melanson EL, Luke AH, Pontzer H, Rood J, Schoeller DA, Westerterp KR, Wong WW; IAEA DLW database group. A standard calculation methodology for human doubly labeled water studies. Cell Rep Med. 2021 Feb 16;2(2):100203. doi: 10.1016/j.xcrm.2021.100203. eCollection 2021 Feb 16. PMID 33665639
- [Background] WEIR JB. New methods for calculating metabolic rate with special reference to protein metabolism. J Physiol. 1949 Aug;109(1-2):1-9. doi: 10.1113/jphysiol.1949.sp004363. No abstract available. PMID 15394301